CLINICAL TRIAL: NCT03441620
Title: Effects of Strawberries on LDL Cholesterol and Insulin Resistance in Overweight/Obese Adults With the Metabolic Syndrome.
Brief Title: The Effects of Strawberries on Blood Cholesterol.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: University of Oklahoma (Other); Oklahoma State University (Other)
Responsible Party: Principal Investigator, Arpita Basu, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1119274
Record Dates: First submitted 2018-02-05; First posted 2018-02-22 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Hyper-LDL-cholesterolemia; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Calorie and fiber-matched control powder
  Interventions: Other: Control powder
- Strawberry one serving (Experimental): Freeze-dried powder equivalent to one serving fresh strawberries per day.
  Interventions: Dietary Supplement: strawberries
- Strawberry two-half servings (Experimental): Freeze-dried powder equivalent to 2.5 serving fresh strawberries per day.
  Interventions: Dietary Supplement: strawberries

INTERVENTIONS:
Dietary Supplement: strawberries — Freeze-dried strawberry powder
  Arms: Strawberry one serving; Strawberry two-half servings
Other: Control powder — Control powder matched for fiber and strawberries
  Arms: Control

SUMMARY:
In this study, we propose to investigate the effects of dietary achievable doses of strawberries on serum LDL-cholesterol (LDL-C) and related lipid profiles, measures of glycemia and insulin resistance, and biomarkers of inflammation in a 14 week controlled crossover study.

DETAILED DESCRIPTION:
The screen visit will involve an 8 hour fasting state and the following procedures:

* Completing screening questionnaire
* Measuring height, weight, blood pressure, and waist size
* Drawing about 30mL blood for blood glucose and lipids and comprehensive metabolic panel All subjects will be asked to follow usual diet and lifestyle, and refrain from other sources of berries and related products while on the study. Subjects will also maintain 3-day food records at screen, 4, 9, and 14 weeks of the study. Height, weight, blood pressure and waist circumference will be measured by trained personnel at MPE 326 (KNS facility for clinical research). Blood draws will be performed by trained phlebotomists (to be hired) at MPE 326, and all procedures will be performed by trained research personnel [PI &Co-PI: Basu, Izuora and graduate student]. In case of blood pressure, an average of at least three readings, 10 min apart, will be measured at each visit for each participant. Blood glucose (fasting and postprandial at two hours) will be determined at each time point. The oral glucose tolerance tests will be conducted at MPE 326 and blood samples will be sent to Quest Diagnostics, Las Vegas. Insulin resistance will be calculated using the homoeostatic model assessment (HOMA-IR). The HOMA-IR is a standard and widely used formula in calculating insulin resistance based on fasting glucose values. Screening and follow-up tests will include clinical laboratory tests for blood glucose, lipids, NMR profiles, C-reactive protein and metabolic panel to determine effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* elevated total and LDL cholesterol (>116 mg/dL)
* body mass index (> or = 30 kg/m2)
* features of the metabolic syndrome

Exclusion Criteria:

* taking glucose and lipid lowering medications (e.g. statins, metformin)
* history of chronic conditions (diabetes, CHD, anemia, renal diseases)
* allergic to strawberries
* pregnant and/or lactating
* smoking
* vegetarian or consuming special diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Serum Lipid profiles | 14 weeks
  Serum LDL, total and HDL cholesterol, triglycerides
Glycemic control | 14 weeks
  Blood glucose
Serum lipid particle concentrations | 14 weeks
  Molar concentrations of serum lipids and particle size
Diabetes control | 14 weeks
  Insulin resistance

SECONDARY OUTCOMES:
Systemic Inflammation | 14 weeks
  Serum C-reactive protein and adipokines
Systemic Anthocyanins | 14 weeks
  Strawberry anthocyanin metabolites measured in serum
Serum metabolomics | 14 weeks
  primary and lipid metabolites in serum

CONTACTS AND LOCATIONS:
Overall Officials: Arpita Basu, PHD, Principal Investigator — University of Nevada at Las Vegas
Locations (3):
- United States (3):
  - University of Nevada at Las Vegas, Las Vegas, Nevada
  - University of Oklahoma Health Sciences Center, OCTSI, Oklahoma City, Oklahoma
  - Oklahoma State University, Stillwater, Oklahoma